CLINICAL TRIAL: NCT06712485
Title: Identification of Biomarkers in Extracellular Vesicles Associated With Marrow Adiposity and Bone Deterioration Caused by Nutritional Deficiencies
Brief Title: Biomarkers in EV Associated With Marrow Adiposity in Anorexia
Acronym: VE_BMAT_AN
Status: Not yet recruiting | Type: Observational
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Sponsor
Other Study IDs: FEIOMM24_001; FEIOMM24_001 (Other Grant/Funding Number: Fundación Española de Investigación Ósea y Metabolismo Mineral)
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-11

CONDITIONS: Anorexia Nervosa Restricting Type; Anorexia Nervosa (DSM-IV Revised Criteria)
Keywords: Extracellular Vesicles; Bone Deterioration; Biomarkers; Bone Marrow Adipose Tissue; Nutritional Deficiencies
MeSH Terms: conditions — Anorexia Nervosa; Malnutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- AN: Patients with Anorexia Nervosa diagnosed according to the DSM-V criteria.
- AN-R: Patients recovered from Anorexia Nervosa
- CON: Healthy subjects of the same age and gender as all other groups

SUMMARY:
The aim of this observational study is to identify biomarkers in extracellular vesicles associated with medullary adiposity occurring in patients with anorexia nervosa. The main question it aims to answer is:

Can this medullary adiposity be associated with the bone deterioration observed in this population?

Participants will be assessed for body composition and a blood sample will be taken by non-invasive techniques.

ELIGIBILITY:
Inclusion Criteria:

For AN group:

* Diagnosis of active AN according to DSM-5 criteria
* BMI of less than 17kg/m2
* Present amenorrhoea in the 3 months prior to the start of the study.

For AN-R group:

* Achieved weight gain of more than 85%.
* Normal menstruation in the last 3 months.

For Control group:

* Population of the same age and gender as the AN and AN-R groups.
* If pubertal population, presenting a chronological age of ± 2 years.
* Normal menstruation
* Normal BMI (>18.5 kg/m2)
* No presence of previous dietary transtrons.

Exclusion Criteria:

* Not receiving oestrogens, contraceptives or glucocorticoids in the 3 months prior to the start of the study.
* Not to suffer from chronic diseases, such as diabetes, pathologies affecting the bone system or thyroid function.
* Do not take calcium or vitamin supplements.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients diagnosed with active anorexia nervosa according to DSM-V criteria (AN group), with a clinical history in the Clinical Management Unit of Endocrinology and Nutrition of the HURS, patients recovered from the disease (AN-R group) and healthy population of the same age and gender as the patients in the previous groups (CON group).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Biomarkers related to medullary adiposity | 1 day
  Blood samples to isolate extracellular vesicles for omics studies

SECONDARY OUTCOMES:
Bone Mineral Density | 1 day
  Bone mineral density measured by densitometry
Body Composition | 1 day
  Fat and muscle mass measured by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Marta Camacho-Cardenosa, pHd, Principal Investigator — Maimonides Biomedical Research Institute of Córdoba
Locations (1):
- Hospital Universitario Reina Sofía, Edificio IMIBIC, Avd. Menedez Pdial, s/n, Córdoba, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Griffith JF, Yeung DK, Ahuja AT, Choy CW, Mei WY, Lam SS, Lam TP, Chen ZY, Leung PC. A study of bone marrow and subcutaneous fatty acid composition in subjects of varying bone mineral density. Bone. 2009 Jun;44(6):1092-6. doi: 10.1016/j.bone.2009.02.022. Epub 2009 Mar 5. PMID 19268721
- [Background] Goto H, Hozumi A, Osaki M, Fukushima T, Sakamoto K, Yonekura A, Tomita M, Furukawa K, Shindo H, Baba H. Primary human bone marrow adipocytes support TNF-alpha-induced osteoclast differentiation and function through RANKL expression. Cytokine. 2011 Dec;56(3):662-8. doi: 10.1016/j.cyto.2011.09.005. Epub 2011 Oct 1. PMID 21963155
- [Background] Ghali O, Al Rassy N, Hardouin P, Chauveau C. Increased Bone Marrow Adiposity in a Context of Energy Deficit: The Tip of the Iceberg? Front Endocrinol (Lausanne). 2016 Sep 16;7:125. doi: 10.3389/fendo.2016.00125. eCollection 2016. PMID 27695438
- [Background] Fazeli PK, Bredella MA, Misra M, Meenaghan E, Rosen CJ, Clemmons DR, Breggia A, Miller KK, Klibanski A. Preadipocyte factor-1 is associated with marrow adiposity and bone mineral density in women with anorexia nervosa. J Clin Endocrinol Metab. 2010 Jan;95(1):407-13. doi: 10.1210/jc.2009-1152. Epub 2009 Oct 22. PMID 19850693
- [Background] Fazeli PK, Bredella MA, Freedman L, Thomas BJ, Breggia A, Meenaghan E, Rosen CJ, Klibanski A. Marrow fat and preadipocyte factor-1 levels decrease with recovery in women with anorexia nervosa. J Bone Miner Res. 2012 Sep;27(9):1864-71. doi: 10.1002/jbmr.1640. PMID 22508185
- [Background] Ambrosi TH, Schulz TJ. The emerging role of bone marrow adipose tissue in bone health and dysfunction. J Mol Med (Berl). 2017 Dec;95(12):1291-1301. doi: 10.1007/s00109-017-1604-7. Epub 2017 Nov 3. PMID 29101431